CLINICAL TRIAL: NCT03550274
Title: A Pilot Study Investigating the Use and Preliminary Effect of the App "Injury-map" in Providing Exercise Rehabilitation for Persons With Acute Lateral Ankle Sprains Seen at the Emergency Department - a Mixed-method Pilot Study
Brief Title: App-based Exercise Intervention for Persons With Acute Ankle Sprain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Copenhagen Center for Health Technology (CACHET) (Unknown); Technical University of Denmark (DTU) (Unknown)
Responsible Party: Principal Investigator, Jonas Bak, Research assistant, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17041467
Record Dates: First submitted 2018-05-01; First posted 2018-06-08 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Ankle Sprains
Keywords: Acute lateral ankle sprain; Acute ankle injury; Ankle sprain; Exercise therapy; App-based rehabilitation; Mixed-method; Pilot Study
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Intervention Model Description: Mixed method pilot cohort study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- App-based exercise rehabilitation (Experimental): Persons with Acute lateral ankle sprain (<48 hours) evaluated by a relevant health specialist in the hospital Emergency Department.
  Interventions: Device: App-based exercise rehabilitation

INTERVENTIONS:
Device: App-based exercise rehabilitation — App-based exercise rehabilitation available on any mobile device and/or tablet using Android or iOS operating systems. The app Injurymap© is hosting the exercise program. The app requires user-registrations and a monthly paid subscription fee to access the exercise program. The participants in this study will not be charged for using the app.
  The exercise program consists of three phases with increasing difficulty. Each phase consists of several categories of exercise types. The categories are 1) mobility, 2) stability/balance, 3) strength and 4) stretching. Within each phase, there can be more than one exercise for each category. This makes it possible to adjust the difficulty of the exercises depending on user-feedback.

SUMMARY:
Acute lateral ankle sprains (ALAS) account for 4-5% of all Emergency Department visits in Denmark. Up to 2/3 of individuals with a history of lateral ankle sprain have prolonged symptoms for several years after their initial injury. Exercise therapy has proven to be a cost-effective rehabilitation in treating ALAS and in preventing re-injury. Injury-map© is an exercise app designed for treating different musculoskeletal problems including ALAS. The app has currently not been tested in a clinical trial with patients suffering from ALAS. This mixed method pilot cohort study aims to investigate the use and preliminary effect of an exercise program on a mobile device in patients with ALAS. The exercise program is designed to be completed within approximately 3 months. However, participants will be followed as long as they complete minimum 1 exercise session per week. If a participant is inactive for two weeks they will be considered completed and contacted for follow-up assessment.

DETAILED DESCRIPTION:
Acute lateral ankle sprains (ALAS) account for 4-5% of all Emergency Department visits in Denmark and is the most common injury in sporting activities. It is often regarded as an innocuous injury but in truth up to 2/3 of individuals with a history of lateral ankle sprain have prolonged symptoms such as pain, decreased function and subjective instability for several years after their initial injury. Exercise therapy has proven to be a cost-effective rehabilitation in treating ALAS and in preventing re-injury. The financial modality of ALAS is high but exercise therapy has proven to be a cost-effective rehabilitation in treating ALAS and in preventing re-injury.

Modern technology has the potential to be a powerful tool in providing easily accessible exercise programs. Injury-map© is an exercise app designed for treating different musculoskeletal problems including ALAS. The exercise program has been developed by health professionals and has the potential to provide an easy-accessible management of ALAS rehabilitation. However, the app has currently not been tested in a clinical trial with patients suffering from ALAS. Before undertaking a large scale trial, the investigators wish to pilot test the app to assess the use and preliminary effect of the app-based exercise program.

This study aims to investigate the use and preliminary effect of an exercise program on a mobile device in patients with ALAS when seen in the Emergency Room at a public hospital. It is designed as a mixed method pilot cohort study. The SPIRIT checklist for trial protocols and the PREPARE trial guide have been used for the overall framework of this protocol.

Approximately 60 participants will be recruited from the Emergency Department (ED) at Hvidovre Hospital (HvH). Health specialists associated with the ED and responsible for ankle examinations will recruit participants . If a health specialist deems a person eligible, they will deliver a bag containing a rubber band and project description. If a participant is willing to participate in the project, they can contact the study administrator by the contact information in the written material. When contact is established participants will receive a voucher for the app, informed consent and a baseline questionnaire.

The exercise program will be available on any mobile device and/or tablet using Android or iOS. It is expected that patients primarily will exercise mainly at home. Participants will be followed as long as they actively use the exercise app or for a maximum of four months. When a participant has been inactive for more than two weeks, the participants are considered finalized and will be contacted for follow-up assessment.

Participants will receive a weekly SMS string where information of return to activity and subjective feeling of instability will be collected. The SMS string will send ever for four months. At follow-up assessment participants will receive a questionnaire containing questions of their experience with the exercise app. A number of participants will be selected to semi-structured interview to elaborate their user experience with the app. This selection will be based on the participants completion of exercises in the app. AT the ED and in the app system recruitment rates and adherence to the exercise program will be extracted.

Baseline characteristics will be summarized with suitable descriptive statistics.

For the aim of investigating the use of the App, adherence will be presented as the number of exercise sessions completed each week as well as average estimations. The results will be compared to an evidence-based exercise dose. Recruitment rates, retention rates will be presented in suitable descriptive tables. Any harms will be addressed individually.

Intervention outcomes will be summarized and tendencies in treatment effect will be compared with comparable literature, however no formal hypothesis testing will be performed, as the study uses a pilot design. Being an exploratory pilot study, the study is designed with a flat outcome structure with multiple evenly valued outcome measures.

Interviews will be recorded and transcribed verbatim. The data will be analysed using a thematic approach. The data will be coded and recurring phrases or words will be grouped into basic themes. These themes will be clustered into global themes which will be verified by comparison to the coded data [23]. Differences between participants who complete the intervention and those who do not will be discussed.

The enrollment process will start in April 2018 and conclude when 60 participants have been enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Acute lateral ankle sprain (< 48 hours) evaluated by a relevant health specialist in the hospital Emergency department (HvH)

Exclusion Criteria:

* Fracture of the leg or foot (Ottawa rules and/or x-ray)
* Previous surgery in the ankle or as a consequence of the current ankle distortion.
* Other serious injury to the body in relation to the ankle injury incidence.
* Serious illness (terminal patients, RA, Fibromyalgia etc).
* Not having a smartphone or tablet.
* Unable to understand Danish.

Ages: 5 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2019-08-03 (Actual); Study Completion 2019-08-03 (Actual)

PRIMARY OUTCOMES:
Return to work | Four months from ankle injury
  Number of whole days absent from work due to the ankle injury
Return to sport | Four months from ankle injury
  Number of exercise sessions not able to fully attend due to the ankle injury
Re-injuries in the same ankle | Four months from ankle injury
  Total number of re-sprains categorized into two groups. 1) Ankle sprains with no time loss and 2) ankle sprains with time-loss defined as unable to continue current activity and/or unable to participate in work/sport activities the next days because of the ankle.
Subjective feeling of ankle stability | Every week from ankle injury until four months after
  0-10 points, where 0 is completely stable and 10 is very unstable. The participant writes a number within the indicated range that equates to their subjective feeling of stability.
Subjective feeling of recovery | Four months from ankle injury
  Do you feel able to do the same activities on the same level as before the injury. answer: YES or NO.
Recruitment rate: Number of potentially eligible participants at the Emergency Department | From start of recruitment to the minimum of 60 participants has been achieved, but maximum 3 months
  Database search off registered ankle injuries at the Emergency Department in the recruitment period
Recruitment rate: Number of persons contacted by the health specialist for information about the study | From start of recruitment to the minimum of 60 participants has been achieved, but maximum 3 months
  Number of delivered recruitment bags containing project information and rubber bands by the health personel at the Emergency Department.
Recruitment rate: Number of persons willing to participate. | From start of recruitment to the minimum of 60 participants has been achieved, but maximum 3 months
  Number of participants who contacts the project administration for participation in the exercise project.
Recruitment rate: Number of persons commencing the exercise program. | From start of recruitment to two weeks after the minimum of 60 participants has been achieved, but maximum 3 months and two weeks.
  Number of participants included in the project who commence the exercise program.
Retention rate: Number of persons completing follow-up assessment. | Four months from ankle injury
  The number of participants completing the four month follow-up questionnaire of the total number included participants.
Retention rate: Number of sms responded. | Four months from ankle injury
  The number of sms responded of the total number of sms send.
Adherence to exercise program: Number of exercise sessions completed. | Four months from ankle injury
  The number of sessions completed is extracted from the app database.
Adherence to exercise program: Number of weeks with minimum one exercise session. | Four months from ankle injury
  The number of sessions completed in each week is extracted from the app database.

OTHER OUTCOMES:
semi-structured interviews | two weeks after ended intervention but maximum 4 months and two weeks after the initial ankle injury.
  To uncover user experiences with the app-based exercise program.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Bak, MSc, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Copenhagen, Hvidove, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bak J, Thorborg K, Clausen MB, Johannsen FE, Kirk JW, Bandholm T. Using the app "Injurymap" to provide exercise rehabilitation for people with acute lateral ankle sprains seen at the Hospital Emergency Department-A mixed-method pilot study. PLOS Digit Health. 2023 May 15;2(5):e0000221. doi: 10.1371/journal.pdig.0000221. eCollection 2023 May. PMID 37186574